CLINICAL TRIAL: NCT01186081
Title: Comparison of Preoperative and Postoperative Radiotherapy and Capecitabine in Locally Advanced Rectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Jong Hoon Kim / Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMC Rectal Pre Vs Post 2004
Record Dates: First submitted 2010-08-18; First posted 2010-08-23 (Estimated); Last update posted 2010-08-23 (Estimated); Status verified 2010-08

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Preoperative CCRT; Postoperative CCRT; Capecitabine
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Preoperative chemoradiotherapy (Experimental): Preoperative chemoradiotherapy with conventional radiation schedule and oral fluoropyrimidine (capecitabine)
  Interventions: Radiation: Preoperative chemoradiotherapy
- Postoperative chemoradiotherapy (Active Comparator): Postoperative chemoradiotherapy with conventional radiation schedule and oral fluoropyrimidine (capecitabine)
  Interventions: Radiation: Postoperative chemoradiotherapy

INTERVENTIONS:
Radiation: Preoperative chemoradiotherapy — Preoperative chemoradiation with conventional radiotherapy (46 Gy in 23 fractions to the whole pelvis followed by a boost dose of 4 Gy in 2 fractions) and oral fluoropyrimidine (capecitabine 825 mg/m2 twice per day without weekend breaks during whole radiotherapy period)
  Other Names: Preoperative CCRT
  Arms: Preoperative chemoradiotherapy
Radiation: Postoperative chemoradiotherapy — Postoperative radiotherapy with conventional radiation schedule (50 Gy in 25 fractions to the whole pelvis) and oral fluoropyrimidine (capecitabine 825 mg/m2 twice per day without weekend breaks during whole radiotherapy period)
  Other Names: Postoperative CCRT
  Arms: Postoperative chemoradiotherapy

SUMMARY:
Based on the potential advantaged of preoperative chemoradiotherapy and oral fluoropyrimidine, the investigators planned a prospective randomized phase III trial which compares preoperative chemoradiotherapy and postoperative chemoradiotherapy with conventional radiation schedule and oral fluoropyrimidine to establish new standard neo-adjuvant therapy regimen in locally advanced rectal cancer.

DETAILED DESCRIPTION:
Although there have been no confirmative data which favored preoperative chemoradiotherapy, preoperative chemoradiation have many theoretical advantage compared with postoperative one. Preoperative radiotherapy with intensive short course regimen showed significant improvement in local control even with TME, but there has been no large prospective randomized trial which proved the efficacy of preoperative chemoradiotherapy compared with the standard postoperative chemoradiotherapy. Although the final result of the German Trial may give the answer for this question, there has been no randomized controlled trial which investigated the efficacy of preoperative chemoradiotherapy using oral fluoropyrimidine which have many theoretical and clinical advantages mentioned above; the German Trial used 5-day continuous infusion of 5-FU. The investigators think that preoperative chemoradiotherapy with oral capecitabine could be new standard regimen in locally advanced rectal cancer, but this regimen must be compared with the standard postoperative chemoradiotherapy through well designed prospective randomized trial. Based on the potential advantaged of preoperative chemoradiotherapy and oral fluoropyrimidine, the investigators planned prospective randomized phase III trial which compares preoperative chemoradiotherapy and postoperative chemoradiotherapy with conventional radiation schedule and oral fluoropyrimidine to establish new standard neo-adjuvant therapy regimen in locally advanced rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed rectal adenocarcinoma
* Tumor located below 10 cm from the anal verge
* Clinical stage T3 or potentially resectable T4, or N+ on endorectal ultrasonography (EUS) and computed tomography (CT)
* Patients must be > 18 years and < 76 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Adequate bone marrow reserve
* Adequate renal function
* Adequate liver function
* Signed informed consent prior to randomization

Exclusion Criteria:

* Evidence of distant metastasis
* Previous history of chemotherapy or radiotherapy
* History of malignancy during recent 5 years other than skin cancer
* Pregnant or lactating woman
* Familial history of colorectal cancer

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2004-03; Primary Completion 2009-04 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | Three year

SECONDARY OUTCOMES:
Overall survival | Three year
Local relapse-free survival | Three year
Sphincter preservation rate | Three year
Treatment related toxicities | Three year

CONTACTS AND LOCATIONS:
Overall Officials: Jong Hoon Kim, M.D., Ph.D., Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea